CLINICAL TRIAL: NCT00818012
Title: Atrial Electromechanical Interval and Pulse Wave Velocity in the Prediction of Recurrence of Atrial Fibrillation In Patients Undergoing Successful Electrical Cardioversion to Sinus Rhythm
Brief Title: Atrial Electromechanical Interval and Pulse Wave Velocity in the Prediction of Recurrence of Atrial Fibrillation
Acronym: APPRAISE
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Other Study IDs: 08-15050
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; atrial electromechanical interval; direct current cardioversion; pulse wave velocity
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to evaluate the utility of the atrial electromechanical interval and pulse wave velocity in the prediction of recurrence of atrial fibrillation among patients who underwent successful direct current cardioversion for atrial fibrillation.

DETAILED DESCRIPTION:
This will be a prospective cohort study designed to evaluate the value of atrial electromechanical interval and pulse wave velocity in the prediction of recurrence of atrial fibrillation among patients with atrial fibrillation with successful direct-current cardioversion to sinus rhythm.

Should cardioversion be successful, a limited 2D echocardiogram will be done and the following information will be measured: atrial electromechanical interval, left atrial volume, left atrial size, ejection fraction, and maximal A-wave transmitral Doppler flow velocity. The presence of left ventricular hypertrophy and valvular heart disease will be recorded. In addition, baseline clinical information including age, gender, medications, presence of HTN, DM, CAD, stroke, and prior history of atrial fibrillation will be obtained.

Radial artery applanation tonometry and pulse wave analysis will be used to calculate a central aortic pressure and other parameters using commercially available SphygmoCor® system. Central aortic pressures will be obtained immediately following measurement of brachial artery pressures. Patients will be seated for 5 minutes in a quiet room after which time blood pressure will be measured over the brachial artery three times at 5 minute intervals. The mean of the last two measurements will be recorded as representative of the brachial artery pressure. After the last measurement, radial artery pressure waveforms of the same arm will be sampled over 10 seconds with a Millar tonometer and calibrated to the average brachial pressure. Waveforms will be processed with dedicated software (SphygmoCor® version 7, AtCor). The software will be used to calculate an averaged radial artery waveform and to derive a corresponding central aortic pressure. Aortic pressure waveforms will be subjected to further analysis by the SphygmoCor® software to identify the time to the peak/shoulder of the first and second pressure wave components (T1, T2) during systole. The pressure at the peak/shoulder of the first component sill be identified as P1 height (outgoing pressure wave) and the pressure difference between P1 and the maximal pressure during systole (∆P or augmentation) will be identified as the reflected pressure wave occurring during systole. Augmentation index (AIx), defined as the ratio of augmentation to central pulse pressure, will be expressed as the percentage: AIx = (∆P/PP) x 100, where P is pressure and PP is pulse pressure. Pulse pressure amplification (PPA) will be expressed as the ratio of central pulse pressure (CPP) to peripheral (brachial) pulse pressure (PPP): PPA = PPP/CPP

Information will be recorded and the patients will be followed by their respective cardiologists and evaluated for recurrence of atrial fibrillation within 6 months.

Primary endpoint for this study is clinical recurrence of atrial fibrillation or 6 month time frame of sustained maintenance of sinus rhythm whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 19 years of age
* History of atrial fibrillation with successful cardioversion to sinus rhythm
* Informed consent to participate in the study

Exclusion Criteria:

* Failure of cardioversion to sinus rhythm
* Use of anti-arrythmic drug therapy
* Refusal to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Atrial Fibrillation
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2008-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Recurrence of Atrial Fibrillation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Ulveling, MD, Principal Investigator — Creighton University Medical Center
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States